CLINICAL TRIAL: NCT00845078
Title: Prospective Outcomes After Reconstruction and Radiotherapy for Breast Cancer
Status: Withdrawn | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: PRO07120002
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2009-02

CONDITIONS: Breast; Radiotherapy; Aesthetics; Treatment Outcome; Surgical Reconstruction
Keywords: Breast; Radiotherapy; Esthetics; Treatment Outcome; Reconstructive Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Immediate reconstruction followed by radiation therapy
- 2: Radiation therapy followed by delayed reconstruction

SUMMARY:
This study examines the aesthetic outcomes of breast reconstruction after mastectomy for breast cancer in patients who require post-mastectomy radiation treatment. Patients will undergo autologous tissue breast reconstruction either in immediate fashion, prior to radiation treatment, or in delayed fashion, after radiation treatment. Both approaches are acceptable and are practiced clinically. this will be an observational prospective cohort study.

The investigators hypothesize that immediate autologous reconstruction patients who undergo subsequent radiation therapy have equivalent aesthetic outcome when compared to those in whom reconstruction is delayed until after radiation, with the additional benefit of avoiding the psychological side effects of breast amputation.

DETAILED DESCRIPTION:
Neo-adjuvant or adjuvant chemo-radiation remains one of the pillars for breast cancer treatment. (1, 2) Administration of radiation before or after autologous soft tissue reconstruction has being shown to alter the aesthetics of the new breast. (3-7) Currently, the optimal timing for autologous breast reconstruction in patients who need postmastectomy radiotherapy remains in debate between surgeons. (8) Various studies have tried to address this problem. However, most of them have been retrospective studies (3, 7, 9) and the prospective ones have not have enough patients, have mixed population of patients or the radiation protocols have not been normalized. (5, 6, 10)

We hypothesize that immediate autologous reconstruction patients who undergo subsequent radiation therapy have equivalent aesthetic outcome when compared to those in whom reconstruction is delayed until after radiation, with the additional benefit of avoiding the psychological side effects of breast amputation.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer requiring mastectomy and post-mastectomy radiation
* Desire for breast reconstruction after mastectomy

Exclusion Criteria:

* Inflammatory breast cancer
* Age < 18 years old
* No desire for breast reconstruction
* Women without need for postmastectomy radiation

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing mastectomy and radiation for breast cancer, who desire breast reconstruction after mastectomy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-12

PRIMARY OUTCOMES:
Aesthetic breast scores | preoperative, 1 month, 6 months, 12 months, 24 months

SECONDARY OUTCOMES:
Quality of life (SF36) | preoperative, 1 month, 6 months, 12 months, 24 months
Patient Breast aesthetic perception (BR23) | preoperative, 1 month, 6 months, 12 months, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Julio A Clavijo-Alvarez, MD, Principal Investigator — University of Pittsburgh; Michael L Gimbel, MD, Study Director — University of Pittsburgh

REFERENCES:
- [Background] Edsander-Nord A, Brandberg Y, Wickman M. Quality of life, patients' satisfaction, and aesthetic outcome after pedicled or free TRAM flap breast surgery. Plast Reconstr Surg. 2001 Apr 15;107(5):1142-53; discussion 1154-5. doi: 10.1097/00006534-200104150-00007. PMID 11373553
- [Result] Tran NV, Chang DW, Gupta A, Kroll SS, Robb GL. Comparison of immediate and delayed free TRAM flap breast reconstruction in patients receiving postmastectomy radiation therapy. Plast Reconstr Surg. 2001 Jul;108(1):78-82. doi: 10.1097/00006534-200107000-00013. PMID 11420508
- [Result] Tran NV, Evans GR, Kroll SS, Baldwin BJ, Miller MJ, Reece GP, Robb GL. Postoperative adjuvant irradiation: effects on tranverse rectus abdominis muscle flap breast reconstruction. Plast Reconstr Surg. 2000 Aug;106(2):313-7; discussion 318-20. doi: 10.1097/00006534-200008000-00011. PMID 10946929
- [Result] Kroll SS, Robb GL, Reece GP, Miller MJ, Evans GR, Baldwin BJ, Wang B, Schusterman MA. Does prior irradiation increase the risk of total or partial free-flap loss? J Reconstr Microsurg. 1998 May;14(4):263-8. doi: 10.1055/s-2007-1000179. PMID 9618094
- [Result] Kroll SS, Coffey JA Jr, Winn RJ, Schusterman MA. A comparison of factors affecting aesthetic outcomes of TRAM flap breast reconstructions. Plast Reconstr Surg. 1995 Sep;96(4):860-4. doi: 10.1097/00006534-199509001-00015. PMID 7652060